CLINICAL TRIAL: NCT07378501
Title: Translation and Psychometric Validation of the Thai Version of the Pediatric Quality of Recovery Score (Thai-PedsQoR)
Brief Title: Thai Version of the Pediatric Quality of Recovery Score (PedSQoR): Translation and Psychometric Validation Study
Acronym: Thai-PedsQoR
Status: Not yet recruiting | Type: Observational
Sponsor: Mahidol University (Other)
Responsible Party: Sponsor
Other Study IDs: Si 1069/2025
Record Dates: First submitted 2026-01-07; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Pediatric Quality of Recovery
Keywords: Pediatric anesthesia; Postoperative recovery; Patient-reported outcomes; Questionnaire validation; Psychometric validation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric patients undergoing surgery: Pediatric patients undergoing surgery who complete the Thai-PedsQoR questionnaire, either by self-report or proxy-report. No intervention or group comparison is performed.

SUMMARY:
Postoperative recovery in children is a complex, multidimensional process that differs substantially from recovery in adults, encompassing physical comfort, emotional well-being, behavioral changes, and psychosocial functioning. While several validated Quality of Recovery (QoR) instruments are widely used in adult perioperative care, equivalent tools for pediatric populations remain limited, particularly in non-English-speaking settings. The Pediatric Quality of Recovery score (PedSQoR) was recently developed to address this gap by providing a comprehensive, patient- and proxy-reported outcome measure specifically designed for children. However, a culturally adapted and psychometrically validated Thai version of this instrument is currently unavailable.

The primary objective of this study is to translate and culturally adapt the PedSQoR into Thai in accordance with the International Society for Pharmacoeconomics and Outcomes Research (ISPOR) guidelines for patient-reported outcome measures. The secondary objective is to evaluate the psychometric properties of the Thai-PedSQoR, including content validity, construct validity, reliability, and responsiveness, in Thai pediatric surgical patients.

This clinical applied research will be conducted at Siriraj Hospital and will include children aged 2-17 years undergoing elective surgery or procedures requiring anesthesia. The translation process will involve forward and backward translation, expert committee review, and cognitive debriefing with parents and children to ensure conceptual equivalence and cultural appropriateness. Psychometric validation will be performed in a cohort of 130 participants, stratified into proxy-report and self-report groups according to age. The Thai-PedSQoR will be administered on postoperative days 2, 6, and 21, alongside anchor measures including pain and global recovery visual analog scales.

The expected outcome of this study is a reliable and valid Thai version of the PedSQoR that can be used in clinical practice, quality improvement initiatives, and future pediatric perioperative research, supporting patient-centered and value-based pediatric surgical care in Thailand.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 2-17 years undergoing day surgery/intervention or surgery/intervention requiring postoperative hospital admission.
* ASA Physical Status I-III.

Exclusion Criteria:

* Patients or parents/guardians who are unable to communicate in Thai.
* Urgent or emergent surgery.
* Children with significant developmental delay or severe systemic disease that interferes with activities of daily living.
* Parents, guardians, or patients who, in the opinion of the investigator, are unlikely to be available to complete follow-up.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population includes pediatric patients undergoing surgical procedures who are assessed for postoperative recovery using the Thai Pediatric Quality of Recovery questionnaire (Thai-PedsQoR). Depending on the child's age and developmental ability, the questionnaire is completed either by the child (self-report) or by a parent or primary caregiver (proxy-report). Expert participants involved in content validity assessment include healthcare professionals with expertise in pediatric perioperative care and patient-reported outcome measurement.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Successful Translation and Cultural Adaptation of the Thai Pediatric Quality of Recovery Questionnaire (Thai-PedsQoR) | With in 2 months after IRB approval
  Completion of the translation and cultural adaptation process of the Pediatric Quality of Recovery Questionnaire (PedSQoR) into Thai, following the ISPOR guidelines. Successful adaptation is defined as finalized Thai-PedsQoR wording approved by forward translation, backward translation, expert review, and cognitive debriefing, with no unresolved major issues identified.

SECONDARY OUTCOMES:
Internal Consistency of the Thai-PedsQoR | From initial questionnaire administration to repeat assessment within 21 days
  Internal consistency will be evaluated using Cronbach's alpha coefficient, which ranges from 0 to 1, with higher values indicating better internal consistency of the questionnaire items.
Responsiveness of the Thai Pediatric Quality of Recovery Questionnaire (Thai-PedsQoR) | From initial questionnaire administration to repeat assessment within 21 days
  Responsiveness will be assessed by changes in Thai-PedsQoR total scores over time following surgery, with higher scores indicating greater levels of the measured attributes as reported, reflecting changes in postoperative recovery trajectories in pediatric patients..
Item-Level Content Validity Index (I-CVI) of the Thai Pediatric Quality of Recovery Questionnaire (Thai-PedsQoR) | Within 3 months after IRB approval
  Item-level Content Validity Index (I-CVI) calculated as the proportion of experts rating each item of the Thai-PedsQoR as relevant (rating of 3 or 4 on a 4-point relevance scale). I-CVI values range from 0 to 1, with higher values indicating greater item relevance.
Scale-Level Content Validity Index (S-CVI) of the Thai Pediatric Quality of Recovery Questionnaire (Thai-PedsQoR) | Within 3 months after IRB approval
  Scale-level Content Validity Index (S-CVI/Ave) calculated as the average of item-level content validity indices across all items of the Thai-PedsQoR. S-CVI values range from 0 to 1, with higher values indicating better overall content validity of the questionnaire.
Content Validity Ratio (CVR) of the Thai Pediatric Quality of Recovery Questionnaire (Thai-PedsQoR) | Within 3 months after IRB approval
  Content Validity Ratio (CVR) calculated using Lawshe's method based on expert ratings of item essentiality. CVR values range from -1 to +1, with higher values indicating greater expert agreement that an item is essential for assessing pediatric postoperative recovery.

CONTACTS AND LOCATIONS:
Locations (1):
- Siriraj Hospital, Bangkok Noi, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Graydon C, Stricker PA, Kelleher S, et al. Development of the Pediatric Scale for Quality of Recovery (PedSQoR). Anesthesiology. 2025;143(2):275-286.